CLINICAL TRIAL: NCT04187053
Title: Clinical and Microbiologic Outcomes of Adjunctive Antimicrobial Photodynamic Therapy in the Non-surgical Treatment of Peri-implant Disease
Brief Title: Clinical and Microbiologic Outcomes of aPDT in the Non-surgical Treatment of Implant Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Academy of Laser Dentistry (Other)
Responsible Party: Principal Investigator, Jiayin Tan, Periodontics Resident, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-DB-19-0873
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-01

CONDITIONS: DENT IMPLANTS; LASER
Keywords: Dental implants; Laser; Antimicrobial photodynamic therapy; Low level laser therapy; Peri-implant mucositis; Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Sodium Chloride; Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional mechanical therapy with aPDT adjunct (Experimental): Traditional non-surgical mechanical debridement along with antimicrobial photodynamic therapy will be done at implant sites by applying a photosensitizing dye methylene blue (0.1mg/ml) with a disposable syringe from the bottom of pocket in a coronal direction. The dye will be applied topically confined to the epithelialized space surrounding the implant fixture and will not be internalized. After 5 minutes in situ, the surrounding gingival tissues will be irradiated at six sites around the implant using a diode laser with a wavelength of 660nm, providing an energy density of 10 J/site, 100mW power, time equal to 100 seconds. After irradiation, the site will be thoroughly rinsed with saline.
  Interventions: Procedure: Conventional mechanical therapy; Drug: Methylene Blue; Device: Light emitting laser
- Conventional mechanical therapy with sham aPDT treatment (Sham Comparator): Control group will have conventional mechanical instrumentation of implant site with "Sham" aPDT treatment with saline and non-light emitting laser
  Interventions: Procedure: Conventional mechanical therapy; Drug: Saline; Device: Non-light emitting laser

INTERVENTIONS:
Procedure: Conventional mechanical therapy — Both experimental and sham arms will receive the Conventional mechanical therapy
Drug: Saline — Sham group will receive saline as a sham for methylene blue
  Arms: Conventional mechanical therapy with sham aPDT treatment
Drug: Methylene Blue — Experimental arm will receive methylene blue
  Arms: Conventional mechanical therapy with aPDT adjunct
Device: Light emitting laser — Experimental arm will receive Light emitting laser
  Arms: Conventional mechanical therapy with aPDT adjunct
Device: Non-light emitting laser — Sham group will receive Non-light emitting laser
  Arms: Conventional mechanical therapy with sham aPDT treatment

SUMMARY:
The purpose of this study is to compare clinical outcomes (change in bleeding sites (BOP) and probing depth reduction (PPD) after mechanical debridement of implant surfaces at sites exhibiting plaque induced inflammation with or without adjunctive antimicrobial photodynamic therapy (aPDT) and assess the microbiologic profile of plaque samples before and after treatment with or without aPDT samples.

ELIGIBILITY:
Inclusion Criteria:

* at least one implant with peri-implant inflammation that requires non-surgical treatment.
* Peri-implant diseases included are peri-implant mucositis and peri-implantitis

Criteria for diagnosis of peri-implant mucositis or peri-implantitis:

1. Red, swollen gingival tissues surrounding the implant
2. Presence of bleeding and/or suppuration on gentle probing around the implant
3. Increased probing depth compared to probing depth after restoration of the implant (greater than 2mm increase in probing depth)
4. May or may not have progressive bone loss in relation to radiographic bone levels assessed either 1 year following restoration of the implant OR ≥3mm of radiographic bone loss from the implant platform -systemically healthy or with controlled common systemic conditions, such as hypertension, that will not affect wound healing.

Exclusion Criteria:

* current heavy smokers (>10 cigarettes/day)
* have diabetes or other systemic diseases that may comprise healing
* take antibiotics within 3 months before the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiayin Tan, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston School of Dentistry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Started | 30 | 26
Completed | 26 | 19
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment | Total
Number analyzed (Participants) | 30 | 26 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.36 (13.32) | 61.03 (15.16) | 62.82 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 26 | 56
Dental Arch [Count of Participants; unit: Participants]
  Maxillary | 19 | 18 | 37
  Mandibular | 11 | 8 | 19
Position of Implant [Count of Participants; unit: Participants]
  Anterior | 6 | 11 | 17
  Posterior | 24 | 15 | 39
Restoration Suprastructure [Count of Participants; unit: Participants]
  Single Crown | 23 | 21 | 44
  Fixed Partial Denture | 3 | 2 | 5
  Healing Abutment | 1 | 1 | 2
  Overdentures | 3 | 2 | 5
Periodontal Diagnosis [Count of Participants; unit: Participants]
  Gingivitis | 15 | 10 | 25
  Periodontitis | 12 | 13 | 25
  Edentulous | 3 | 3 | 6
Width of Buccal Keratinized gingiva [Mean (Standard Deviation); unit: millimeters] | 2.37 (0.72) | 3.11 (0.86) | 2.71 (.78)

OUTCOME MEASURES:

1. Primary Outcome: Mean Probing Pocket Depth
Description: Periodontal pocket depth was measured from the free gingival margin to the base of the pocket, with a UNC periodontal probe with 1mm measurement units. It was assessed at 6 sites per implant: mesiobuccal, mid-buccal, distobuccal, distolingual, mid-lingual, and mesiolingual. For each participant, an average of the depths of the 6 sites is reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 26
millimeters | 4.62 (0.49) | 4.45 (0.70)

2. Primary Outcome: Mean Probing Pocket Depth
Description: as for outcome 1
Time Frame: 6 weeks post treatment
Population: Data were not collected for 4 participants in the Conventional mechanical therapy with aPDT adjunct arm. Data were not collected for 7 participants in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 26 | 19
millimeters | 3.92 (0.63) | 3.54 (0.74)

3. Primary Outcome: Mean Probing Pocket Depth
Description: as for outcome 1
Time Frame: 12 weeks post treatment
Population: Data were not collected for 1 participant in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 25
millimeters | 4.02 (0.66) | 3.63 (0.59)

4. Primary Outcome: Improvement in Sites as Indicated by Reduction in Inflammation as Assessed by Clinical Attachment Loss
Time Frame: Baseline
Population: Data were not collected for this outcome measure
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Improvement in Sites as Indicated by Reduction in Inflammation as Assessed by Clinical Attachment Loss
Time Frame: 6 weeks post treatment
Population: Data were not collected for this outcome measure
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Improvement in Sites as Indicated by Reduction in Inflammation as Assessed by Clinical Attachment Loss
Time Frame: 12 weeks post treatment
Population: Data were not collected for this outcome measure
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Number of Bleeding Sites Per Participant as Assessed by Bleeding on Probing
Description: Bleeding on probing (BOP) will be assessed, where each of 6 gingival areas (mesiobuccal, mid-buccal, distobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be gently swept by the periodontal probe just within the gingival sulcus of the implant and the presence or absence of bleeding will be recorded.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Bleeding sites
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 26
Bleeding sites | 4.42 (0.85) | 3.53 (0.79)

8. Primary Outcome: Number of Bleeding Sites Per Participant as Assessed by Bleeding on Probing
Description: as for outcome 7
Time Frame: 6 weeks post treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Bleeding sites
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 26 | 19
Bleeding sites | 3.11 (1.21) | 2.13 (1.29)

9. Primary Outcome: Number of Bleeding Sites Per Participant as Assessed by Bleeding on Probing
Description: as for outcome 7
Time Frame: 12 weeks post treatment
Population: Data were not collected for 1 participant in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: Bleeding sites
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 25
Bleeding sites | 3.2 (0.85) | 2.51 (1.04)

10. Primary Outcome: Number of Sites With Plaque Per Participant
Description: Presence of plaque was evaluated at six sites (mesiobuccal, mid-buccal, distobuccal, distolingual, mid-lingual, and mesiolingual) around the implant surface and the presence of plaque will be recorded.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: sites with plaque
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 26
sites with plaque | 4.06 (0.95) | 4.07 (1.06)

11. Primary Outcome: Number of Sites With Plaque Per Participant
Description: as for outcome 10
Time Frame: 6 weeks post treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: sites with plaque
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 26 | 19
sites with plaque | 3.19 (1.42) | 2.86 (1.72)

12. Primary Outcome: Number of Sites With Plaque Per Participant
Description: as for outcome 10
Time Frame: 12 weeks post treatment
Population: Data were not collected for 1 participant in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: sites with plaque
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 25
sites with plaque | 3.13 (1.07) | 3.12 (1.09)

13. Primary Outcome: Max Probing Pocket Depth
Description: Periodontal pocket depth was measured from the free gingival margin to the base of the pocket, with a UNC periodontal probe with 1mm measurement units. It was assessed at 6 sites per implant: mesiobuccal, mid-buccal, distobuccal, distolingual, mid-lingual, and mesiolingual. For each participant, the depth of the deepest of the 6 sites is reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 26
millimeters | 6.16 (0.75) | 6.34 (1.31)

14. Primary Outcome: Max Probing Pocket Depth
Description: as for outcome 13
Time Frame: 6 weeks post treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 26 | 19
millimeters | 5.23 (1.00) | 4.16 (1.23)

15. Primary Outcome: Max Probing Pocket Depth
Description: as for outcome 13
Time Frame: 12 weeks post treatment
Population: Data were not collected for 1 participant in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 30 | 25
millimeters | 5.53 (0.95) | 4.76 (0.86)

16. Secondary Outcome: Alpha Diversity as Indicated by Analysis of 16S rRNA Gene Data From Plaque Samples
Description: Plaque samples will be taken from the deepest probing site of each implant at baseline and 12 weeks after aPDT. To assess bacteria in the sample, the V4 region of the 16S rRNA gene will be PCR amplified and sequenced, and 16S rRNA gene data will then be analyzed to determine the alpha diversity of the microbiota community at the implant site. In this study, the minimum alpha diversity is 1 and the maximum is 2501. A higher alpha diversity indicates a higher number of bacterial or taxonomic "units" in the sample.
Time Frame: Baseline
Population: Data were not collected for 13 participants in the Conventional mechanical therapy with aPDT adjunct arm. Data were not collected for 10 participants in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: Observed Taxonomic Units (OTUs)
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 17 | 16
Observed Taxonomic Units (OTUs) | 100.98 (22.53) | 92.74 (30.06)

17. Secondary Outcome: Alpha Diversity as Indicated by Analysis of 16S rRNA Gene Data From Plaque Samples
Description: as for outcome 16
Time Frame: 12 weeks post treatment
Population: Data were not collected for 10 participants in the Conventional mechanical therapy with aPDT adjunct arm. Data were not collected for 11 participants in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: Observed Taxonomic Units (OTUs)
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 20 | 15
Observed Taxonomic Units (OTUs) | 105.11 (29.92) | 88.68 (25.65)

18. Secondary Outcome: Levels of Immunologic Biomarkers in Peri-implant Sulcular Fluid (PISF) Sample as Assessed by Multiplexed Fluorescent Bead-based Immunoassay
Description: PISF samples will be taken from six sites of each implant at baseline and 12 weeks after aPDT. The levels of interleukin IL-1a, IL-1b, IL-6, IL-8, IL-10, IL-12, IL-7A, tumor necrosis factor (TNF)-a, C-reactive protein, osteoprotegerin, leptin, and adiponectin will be determined using multiplex proteomic immunoassays.
Time Frame: Baseline
Population: Samples were not tested for the presence of IL-7A, C-reactive protein, osteoprotegerin, leptin and adiponectin. Data were not collected for 24 participants in the Conventional mechanical therapy with aPDT adjunct arm. Data were not collected for 22 participants in the Conventional mechanical therapy with sham aPDT treatment arm.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 6 | 4
picograms per milliliter
  IL-1alpha | 74.13 (56.69) | 42.49 (5.65)
  IL-1beta | 391.24 (451.39) | 324.87 (415.13)
  IL-6 | 26.05 (24.10) | 39.88 (58.02)
  IL-8 | 1283.36 (1094.82) | 1134.66 (950.49)
  IL-10 | 3.20 (1.04) | 2.37 (1.01)
  IL-12 | 1.30 (0.18) | 1.37 (0.28)
  IL-7A: number analyzed (Participants) | 0 | 0
  tumor necrosis factor (TNF)-alpha | 4.06 (2.187) | 3.82 (1.89)
  C-reactive protein: number analyzed (Participants) | 0 | 0
  osteoprotegerin: number analyzed (Participants) | 0 | 0
  leptin: number analyzed (Participants) | 0 | 0
  adiponectin: number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Levels of Immunologic Biomarkers in Peri-implant Sulcular Fluid (PISF) Sample as Assessed by Multiplexed Fluorescent Bead-based Immunoassay
Description: as for outcome 18
Time Frame: 12 weeks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
Number analyzed (Participants) | 6 | 4
picograms per milliliter
  IL-1alpha | 97.91 (52.63) | 94.97 (40.14)
  IL-1beta | 444.11 (478.65) | 177.13 (174.70)
  IL-6 | 24.43 (16.32) | 25.33 (31.99)
  IL-8 | 1691.34 (1411.79) | 1478.70 (1908.61)
  IL-10 | 10.65 (11.28) | 3.17 (2.53)
  IL-12 | 1.33 (0.18) | 1.30 (0.14)
  IL-7A: number analyzed (Participants) | 0 | 0
  tumor necrosis factor (TNF)-alpha | 4.53 (2.46) | 3.52 (0.46)
  C-reactive protein: number analyzed (Participants) | 0 | 0
  osteoprotegerin: number analyzed (Participants) | 0 | 0
  leptin: number analyzed (Participants) | 0 | 0
  adiponectin: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Conventional Mechanical Therapy With aPDT Adjunct | Conventional Mechanical Therapy With Sham aPDT Treatment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/26
Other Adverse Events (participants affected / at risk) | 0/30 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT04187053/Prot_SAP_000.pdf